CLINICAL TRIAL: NCT01106586
Title: A Phase 3, Randomized, Double-Blind Study to Evaluate the Safety and Efficacy of Elvitegravir/Emtricitabine/Tenofovir Disoproxil Fumarate/GS-9350 Versus Ritonavir-Boosted Atazanavir Plus Emtricitabine/Tenofovir Disoproxil Fumarate in HIV-1 Infected, Antiretroviral Treatment-Naive Adults
Brief Title: Study to Evaluate the Safety and Efficacy of Stribild Versus Ritonavir-Boosted Atazanavir Plus Truvada in Human Immunodeficiency Virus, Type 1 (HIV-1) Infected, Antiretroviral Treatment-Naive Adults
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GS-US-236-0103
Record Dates: First submitted 2010-04-14; First posted 2010-04-20 (Estimated); Results first posted 2012-10-22 (Estimated); Last update posted 2015-11-11 (Estimated); Status verified 2015-10

CONDITIONS: HIV; HIV Infections
Keywords: HIV 1 Infection; Treatment Naive
MeSH Terms: conditions — HIV Infections | interventions — Elvitegravir, Cobicistat, Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination; Ritonavir; Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Stribild (Experimental)
  Interventions: Drug: Stribild; Drug: ATV Placebo; Drug: RTV Placebo; Drug: FTC/TDF Placebo
- ATV/r + FTC/TDF (Active Comparator)
  Interventions: Drug: ATV; Drug: Ritonavir; Drug: FTC/TDF; Drug: Stribild Placebo

INTERVENTIONS:
Drug: Stribild — Stribild (EVG 150 mg/COBI 150 mg/FTC 200 mg/TDF 300 mg) STR administered orally once daily
  Arms: Stribild
Drug: ATV — Atazanavir 300 mg capsule administered orally once daily
  Arms: ATV/r + FTC/TDF
Drug: Ritonavir — Ritonavir (RTV; /r) 100 mg tablet administered orally once daily
  Other Names: Norvir®
  Arms: ATV/r + FTC/TDF
Drug: FTC/TDF — FTC/TDF 200/300 mg tablet administered orally once daily
  Other Names: Truvada
  Arms: ATV/r + FTC/TDF
Drug: Stribild Placebo — Placebo to match Stribild administered orally once daily
  Arms: ATV/r + FTC/TDF
Drug: ATV Placebo — Placebo to match ATV administered orally once daily
  Arms: Stribild
Drug: RTV Placebo — Placebo to match RTV administered orally once daily
  Arms: Stribild
Drug: FTC/TDF Placebo — Placebo to match FTC/TDF administered orally once daily
  Arms: Stribild

SUMMARY:
To evaluate the safety and efficacy of Stribild®, a single tablet regimen (STR) containing fixed doses of elvitegravir (EVG)/cobicistat (COBI [GS-9350])/emtricitabine (FTC)/tenofovir disoproxil fumarate (TDF) versus ritonavir-boosted atazanavir (ATV/r) plus the standard of care nucleoside reverse transcriptase inhibitor (NRTI) backbone FTC/TDF (Truvada®). ATV/r + FTC/TDF was selected as the active comparator for this study as it is a preferred protease inhibitor-based regimen in guidelines for the treatment of HIV-1 infected, antiretroviral treatment-naive adults.

ELIGIBILITY:
Inclusion Criteria:

* Ability to understand and sign a written informed consent form, which must be obtained prior to initiation of study procedures
* Plasma HIV-1 RNA levels ≥ 5,000 copies/mL at screening
* No prior use of any approved or investigational antiretroviral drug for any length of time
* Screening genotype report must show sensitivity to FTC, TDF, and ATV
* Normal electrocardiogram (ECG)
* Adequate renal function (estimated glomerular filtration rate ≥ 70 mL/min according to the Cockcroft Gault formula)
* Hepatic transaminases (aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 5 x the upper limit of the normal range (ULN)
* Total bilirubin ≤ 1.5 mg/dL, or normal direct bilirubin
* Adequate hematologic function
* Serum amylase ≤ 5 x ULN
* Males and Females of childbearing potential must agree to utilize highly effective contraception methods from screening throughout the duration of study treatment and for 30 days following the last dose of study drug
* Age ≥ 18 years
* Life expectancy ≥ 1 year

Exclusion Criteria:

* A new acquired immunodeficiency syndrome (AIDS)-defining condition diagnosed within the 30 days prior to screening
* Receiving drug treatment for hepatitis C, or anticipated to receive treatment for hepatitis C
* Subjects experiencing decompensated cirrhosis
* Females who are breastfeeding
* Positive serum pregnancy test (female of childbearing potential)
* Implanted defibrillator or pacemaker
* Current alcohol or substance use judged by the Investigator to potentially interfere with subject study compliance
* History of malignancy within the past 5 years or ongoing malignancy other than cutaneous Kaposi's sarcoma, basal cell carcinoma, or resected, noninvasive cutaneous squamous carcinoma
* Active, serious infections (other than HIV-1 infection) requiring parenteral antibiotic or antifungal therapy within 30 days prior to baseline
* Medications contraindicated for use with EVG, COBI, FTC, TDF, ATV, or ritonavir or subjects with any known allergies to the excipients of Stribild tablets, Truvada tablets, ATV capsules or ritonavir tablets
* Participation in any other clinical trial without prior approval
* Any other clinical condition or prior therapy that, in the opinion of the Investigator, would make the subject unsuitable for the study or unable to comply with the dosing requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 708 (Actual)
Dates: Start 2010-04; Primary Completion 2011-09 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marshall Fordyce, MD, Study Director — Gilead Sciences
Locations (146):
- United States (86):
  - Spectrum Medical Group, Phoenix, Arizona
  - Health for Life Clinic PLLC, Little Rock, Arkansas
  - AHF Research Center, Beverly Hills, California
  - CSI Clinical Trials, Inc., Costa Mesa, California
  - Apex Research, LLC, Denver, California
  - Kaiser Permanente Hospital, Hayward, California
  - Living Hope Clinical Foundation, Long Beach, California
  - Kaiser Permanente, Los Angeles, California
  - Los Angeles Gay and Lesbian Center DBA Jeffrey Goodman Special Care Clinic, Los Angeles, California
  - Peter J Ruane, MD, Inc, Los Angeles, California
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Anthony Mills MD Inc, Los Angeles, California
  - Orange Coast Medical Group, Newport Beach, California
  - Alameda County Medical Center, Oakland, California
  - East Bay AIDS Center, Oakland, California
  - Stanford University, Palo Alto, California
  - University of California, Davis Medical Center, Sacramento, California
  - Kaiser Permanente Medical Group, Sacramento, California
  - La Playa Medical Group and Clinical Research, San Diego, California
  - Metropolitan Medical, San Francisco, California
  - Kaiser Permanente Medical Center, Clinical Trials Unit, San Francisco, California
  - National Jewish Health, Denver, Colorado
  - Yale University HIV Clinical Trials Program, New Haven, Connecticut
  - The Stamford Hospital, Stamford, Connecticut
  - Dupont Circle Physicians Group, Washington D.C., District of Columbia
  - Whitman Walker Clinic, Washington D.C., District of Columbia
  - Capital Medical Associates, PC, Washington D.C., District of Columbia
  - George Washington University Medical Faculty Associates, Washington D.C., District of Columbia
  - Therafirst Medical Center, Fort Lauderdale, Florida
  - Broward Health/Comprehensive Care Center, Fort Lauderdale, Florida
  - Gary J. Richmond,M.D., P.A., Fort Lauderdale, Florida
  - Midway Immunology and Research Center, Ft. Pierce, Florida
  - The Kinder Medical Group, Miami, Florida
  - Wohlfeiler, Piperato and Associates, LLC, Miami Beach, Florida
  - Orlando Immunology Center, Orlando, Florida
  - IDOCF/ ValueHealthMD, LLC, Orlando, Florida
  - University of South Florida HIV Clinical Research Unit / Hillsborough County Health Department, Tampa, Florida
  - Infectious Disease Research Institute Inc., Tampa, Florida
  - St. Joseph's Comprehensive Research Institute, Tampa, Florida
  - Treasure Coast Infectious Disease Consultants, Vero Beach, Florida
  - AIDS Research Consortium of Atlanta, Atlanta, Georgia
  - Infectious Disease Solutions, PC, Atlanta, Georgia
  - Mercer University School of Medicine, Macon, Georgia
  - Leahi Hospital, Honolulu, Hawaii
  - Ruth M. Rothstein CORE Center, Chicago, Illinois
  - Howard Brown Health Center, Chicago, Illinois
  - The Research Institute, Springfield, Massachusetts
  - Baystate Infectious Diseases Clinical Research, Springfield, Massachusetts
  - Be Well Medical Center, Berkley, Michigan
  - Henry Ford Health System, Detroit, Michigan
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - CentralWest Clinical Research, St Louis, Missouri
  - Division of Infectious Diseases, St. Louis University Medical Center, St Louis, Missouri
  - Southampton Healthcare, St Louis, Missouri
  - ID Care, Hillsborough, New Jersey
  - Saint Michaels Medical Center, Newark, New Jersey
  - South Jersey Infectious Disease, Somers Point, New Jersey
  - Garden State Infectious Diseases Associates, PA, Voorhees Township, New Jersey
  - Upstate ID Association, Albany, New York
  - Albany Medical College, Albany, New York
  - STAR Health Care Center (SUNY Downstate), Brooklyn, New York
  - North Shore University Hospital, Manhasset, New York
  - Greiger Clinic, Mount Vernon, New York
  - Beth Israel Medical Center, New York, New York
  - Chelsea Village Medical, PC, New York, New York
  - AIDS Care, Rochester, New York
  - Montiefiore Medical Center- AIDS Center, The Bronx, New York
  - Carolinas Medical Center-Myers Park, Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - East Carolina University, Greenville, North Carolina
  - Rosedale Infectious Diseases, Huntersville, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Summa Health System, Akron, Ohio
  - Division of Infectious Diseases, Thomas Jefferson University, Philadelphia, Pennsylvania
  - Philadelphia FIGHT, Philadelphia, Pennsylvania
  - University of South Carolina, Columbia, South Carolina
  - Nicholaos C. Bellos, MD, PA (Southwest Infectious Disease Clinical Research, Inc.), Dallas, Texas
  - Trinity Health and Wellness Center/AIDS Arms, Inc., Dallas, Texas
  - Tarrant County Infectious Disease Associates, Fort Worth, Texas
  - Garcia's Family Health Group, Harlingen, Texas
  - Dr. Joseph C. Gathe MD (Therapeutic Concepts, PA), Houston, Texas
  - Gordon E. Crofoot MD PA, Houston, Texas
  - Research Access Network, Houston, Texas
  - DCOL Center for Clinical Research, Longview, Texas
  - Clinical Alliance for Research & Education, Infectious Diseases (CARE-ID), Annandale, Virginia
  - Peter Shalit, M.D., Seattle, Washington
- Australia (8):
  - Holdsworth House Medical practice, Darlinghurst, New South Wales
  - National Centre in HIV Epidemiology and Clinical Research (NCHECR), University of New South Wales, Darlinghurst, New South Wales
  - Albion Street Centre, Sydney, New South Wales
  - East Sydney Doctors, Sydney, New South Wales
  - Melbourne Health - Royal Melbourne Hospital Campus (Sexual Health Clinic), Carlton, Victoria
  - Alfred Hospital, Melbourne, Victoria
  - Northside Clinic, Melbourne, Victoria
  - Taylor Square Private Clinica, Darlinghurst
- Austria (3):
  - LKH Graz West, Graz
  - Department of Dermatology, Division of Immunology, Allergy & Inf. Diseases; Medical University Vienna, Vienna
  - Interne Lungenabteilung, SMZ Baumgartner Hoehe - Otto-Wagner-Spital, Vienna
- Belgium (3):
  - CHU Saint-Pierre University Hospital, Brussels
  - Hôpital Universitaire Erasme - ULB, Brussels
  - University of Ghent, Ghent
- Canada (7):
  - Southern Alberta Clinic, Calgary, Alberta
  - Winnipeg Regional Health Authority - Health Sciences Centre Winnipeg, Winnipeg, Manitoba
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - Canadian Immunodeficiency Research Collaborative (CIRC) Inc., Toronto, Ontario
  - University Health Network, Toronto General Hospital, Toronto, Ontario
  - Clinique medicale l'Actuel, Montreal, Quebec
  - Clinique Medicale du Quartier Latin, Montreal, Quebec
- Epidemiklinikken 5112, Rigshospitalet, Copenhagen, Denmark
- France (11):
  - Service des Maladies Infectieuses, CHU de Caen, Caen
  - Hôpital de la Croix Rousse - Maladies Infectieuses et Tropicales, Lyon
  - CHU Gui de Chauliac, Maladies Infectieuses Dpt, Montpellier
  - CHU de Nantes Hopital de l'Hotel Dieu, Nantes
  - Centre Hospitalier Universitaire de Nice, Nice
  - Department of Infectious Diseases, Saint-Louis hospital, Paris
  - Hopital Saint Antoine, Service De Maladies Infectieuses, Paris
  - Bichat Hospital, Paris
  - Tenon Hospital, UPMC, Paris
  - Hopital Pitie-Salpetriere, Paris
  - Centre Hospitalier de Tourcoing, Tourcoing
- Germany (8):
  - University of Bonn, Dep. of Internal Medicine I, HIV-Outpatient Clinic, Bonn
  - University of Cologne, Department of Internal Medicine, Cologne
  - Center for HIV and Hepatogastroenterology, Düsseldorf
  - Infektio Research GmbH / Infektiologikum Frankfurt, Frankfurt am Main
  - Klinikum der Goethe-Universitaet, Medizinische Klinik II, Schwerpunkt HIV, Haus 68, Frankfurt am Main
  - ICH Study Center Hamburg, Hamburg
  - University Medical Center Hamburg-Eppendorf, Infectious Diseases Unit, Hamburg
  - MUC Research GmbH, München
- Italy (3):
  - Fondazione Centro San Raffaele del Monte Tabor, Milan
  - National Institute for Infectious Diseases "L. Spallanzani" IRCCS, Rome
  - Dipartimento di Malattie Infettive, Torino
- Unidad de VIH, Hospital Civil de Guadalajara, Fray Antonio Alcalde, Guadalajara, Jalisco, Mexico
- Netherlands (2):
  - Onze lieve vrouw gasthuis, Amsterdam
  - Erasmus MC, Internal Medicine, Section of Infectious Diseases, Rotterdam
- Serviço de Doenças Infecciosas, Hospital de São João, Porto, Portugal
- Puerto Rico (2):
  - Clinical Research Puerto Rico, San Juan
  - VA Caribbean Healthcare System, San Juan
- Venhälsan, Södersjukhuset, Stockholm, Sweden
- CHUV, Lausanne, Canton of Vaud, Switzerland
- Thailand (2):
  - Ramathibodi Hospital, Mahidol University, Bangkok
  - Siriraj Hospital, Bangkok
- United Kingdom (6):
  - Brighton and Sussex University Hospitals NHS Trust, Brighton, East Sussex
  - North Manchester General Hospital, Manchester, Lancashire
  - Barts and the London NHS Trust, London
  - Homerton University Hospital, London
  - Chelsea and Westminster Hospital Foundation Trust, London
  - St. Mary's Hospital, London (Imperial College, London), London

REFERENCES:
- [Result] DeJesus E, Rockstroh JK, Henry K, Molina JM, Gathe J, Ramanathan S, Wei X, Yale K, Szwarcberg J, White K, Cheng AK, Kearney BP; GS-236-0103 Study Team. Co-formulated elvitegravir, cobicistat, emtricitabine, and tenofovir disoproxil fumarate versus ritonavir-boosted atazanavir plus co-formulated emtricitabine and tenofovir disoproxil fumarate for initial treatment of HIV-1 infection: a randomised, double-blind, phase 3, non-inferiority trial. Lancet. 2012 Jun 30;379(9835):2429-2438. doi: 10.1016/S0140-6736(12)60918-0. PMID 22748590
- [Result] Rockstroh JK, DeJesus E, Henry K, Molina JM, Gathe J, Ramanathan S, Wei X, Plummer A, Abram M, Cheng AK, Fordyce MW, Szwarcberg J; GS-236-0103 Study Team. A randomized, double-blind comparison of coformulated elvitegravir/cobicistat/emtricitabine/tenofovir DF vs ritonavir-boosted atazanavir plus coformulated emtricitabine and tenofovir DF for initial treatment of HIV-1 infection: analysis of week 96 results. J Acquir Immune Defic Syndr. 2013 Apr 15;62(5):483-6. doi: 10.1097/QAI.0b013e318286415c. PMID 23337366
- [Result] Clumeck N, Molina JM, Henry K, Gathe J, Rockstroh JK, DeJesus E, Wei X, White K, Fordyce MW, Rhee MS, Szwarcberg J; GS-236-0103 Study Team. A randomized, double-blind comparison of single-tablet regimen elvitegravir/cobicistat/emtricitabine/tenofovir DF vs ritonavir-boosted atazanavir plus emtricitabine/tenofovir DF for initial treatment of HIV-1 infection: analysis of week 144 results. J Acquir Immune Defic Syndr. 2014 Mar 1;65(3):e121-4. doi: 10.1097/QAI.0000000000000089. No abstract available. PMID 24346640

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at 146 sites in 16 countries. The first participant was screened on 06 April 2010. The last study visit occurred on 18 September 2014.
Pre-assignment Details: 1017 subjects were screened.
Groups:
- Stribild: Stribild® (elvitegravir (EVG) 150 mg/cobicistat (COBI) 150 mg/emtricitabine (FTC) 200 mg/tenofovir disoproxil fumarate (TDF) 300 mg) plus placebo to match atazanavir/ritonavir (ATV/r) + FTC/TDF once daily
- ATV/r + FTC/TDF: ATV/r 300/100 mg tablet plus FTC 200 mg/TDF 300 mg tablet plus placebo to match Stribild once daily
Period: Overall Study
Arm/Group | Stribild | ATV/r + FTC/TDF
Started | 353 | 355
Completed | 68 | 70
Not Completed | 285 | 285
Not completed — Adverse Event | 9 | 15
Not completed — Death | 1 | 3
Not completed — Pregnancy | 2 | 2
Not completed — Lack of Efficacy | 1 | 0
Not completed — Investigator's Discretion | 5 | 8
Not completed — Withdrew Consent | 18 | 30
Not completed — Lost to Follow-up | 24 | 20
Not completed — Participant Noncompliance | 12 | 10
Not completed — Protocol Violation | 1 | 0
Not completed — Participant Transferred to Another Study | 212 | 197

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set: participants who were randomized into the study and received at least 1 dose of study drug
Groups:
- Stribild: Stribild (EVG 150 mg/COBI 150 mg/FTC 200 mg/TDF 300 mg) plus placebo to match ATV/r + FTC/TDF once daily
- Total: Total of all reporting groups
Arm/Group | Stribild | ATV/r + FTC/TDF | Total
Number analyzed (Participants) | 353 | 355 | 708
Age, Continuous [Mean (Standard Deviation); unit: years] | 38 (10.5) | 39 (9.8) | 38 (10.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 39 | 68
  Male | 324 | 316 | 640
Race/Ethnicity, Customized [Number; unit: participants]
  American Indian or Alaska Native | 2 | 3 | 5
  Asian | 17 | 17 | 34
  Black or African Heritage | 72 | 47 | 119
  Native Hawaiian or Pacific Islander | 1 | 2 | 3
  White | 250 | 277 | 527
  Other | 11 | 9 | 20
Region of Enrollment [Number; unit: participants]
  Portugal | 1 | 2 | 3
  United States | 197 | 185 | 382
  Thailand | 7 | 4 | 11
  Austria | 12 | 8 | 20
  United Kingdom | 11 | 15 | 26
  Switzerland | 0 | 2 | 2
  Italy | 9 | 5 | 14
  France | 23 | 23 | 46
  Mexico | 3 | 2 | 5
  Canada | 19 | 22 | 41
  Belgium | 9 | 12 | 21
  Australia | 30 | 32 | 62
  Denmark | 1 | 2 | 3
  Netherlands | 2 | 4 | 6
  Germany | 29 | 36 | 65
  Sweden | 0 | 1 | 1
HIV Disease Status [Number; unit: participants]
  Asymptomatic | 285 | 293 | 578
  Symptomatic HIV Infections | 36 | 38 | 74
  AIDS | 32 | 24 | 56
Hepatitis B Virus (HBV) Infection Status [Number; unit: participants]
  Negative | 347 | 346 | 693
  Positive | 5 | 7 | 12
  Indeterminate | 0 | 1 | 1
  Not done | 1 | 1 | 2
Hepatitis C Virus (HCV) Infection Status [Number; unit: participants]
  Negative | 335 | 344 | 679
  Positive | 18 | 10 | 28
  Indeterminate | 0 | 0 | 0
  Not done | 0 | 1 | 1
HIV-1 RNA Category (copies/mL) [Number; unit: participants]
  ≤ 100,000 copies/mL | 203 | 214 | 417
  > 100,000 copies/mL | 150 | 141 | 291
CD4 Cell Count (/µL) [Number; unit: participants]
  ≤ 50 μL | 12 | 5 | 17
  51 to ≤ 200 μL | 42 | 34 | 76
  201 to ≤ 350 μL | 122 | 124 | 246
  351 to ≤ 500 μL | 122 | 122 | 244
  > 500 μL | 55 | 70 | 125

OUTCOME MEASURES:

1. Primary Outcome: The Percentage of Participants With Virologic Success Using the Food and Drug Administration (FDA)-Defined Snapshot Analysis as Determined by the Achievement of HIV-1 Ribonucleic Acid (RNA) < 50 Copies/mL at Week 48
Time Frame: Week 48
Population: ITT analysis set: participants who were randomized into the study and received at least 1 dose of study drug
Measure: Number; unit: percentage of participants
Arm/Group | Stribild | ATV/r + FTC/TDF
Number analyzed (Participants) | 353 | 355
percentage of participants | 89.5 | 86.8
Statistical Analysis 1: Comparison: Stribild vs ATV/r + FTC/TDF; The null hypothesis was that the Stribild group is at least 12% worse than the ATV/r + Truvada group with respect to percentage of participants achieving HIV-1 RNA < 50 copies/mL (response rate as defined by the snapshot analysis algorithm) at Week 48; the alternative hypothesis was that the response rate in the Stribild group is less than 12% worse than that in the ATV/r + Truvada Group; Test type: Non-Inferiority or Equivalence — A total of 700 HIV-1 infected participants, randomized in a 1:1 ratio to 2 groups would achieve at least 95% power to establish noninferiority in Week 48 response (HIV-1 RNA < 50 copies/mL per the FDA-defined snapshot analysis) rate difference between the 2 groups. For sample size and power computation, it was assumed that both treatment groups have a response rate of 0.795, a noninferiority margin of 0.12, and that the significance level of the test is at a one-sided, 0.025 level; Difference in response rates = 3.0, 95.2% CI 2-sided [-1.9 to 7.8] — To preserve the overall alpha level: 0.05, accounting for 2 interim analyses for Independent Data Monitoring Committee meetings, the 95.2% CI was computed using normal approximation stratified by baseline HIV-1 RNA (≤ 100,000 or > 100,000 copies/mL)

2. Secondary Outcome: The Percentage of Participants With Virologic Success Using the FDA-Defined Snapshot Analysis as Determined by the Achievement of HIV-1 RNA < 50 Copies/mL at Week 96
Time Frame: Week 96
Population: ITT Analysis Set
Measure: Number; unit: percentage of participants
Arm/Group | Stribild | ATV/r + FTC/TDF
Number analyzed (Participants) | 353 | 355
percentage of participants | 83.3 | 82.3

3. Secondary Outcome: The Percentage of Participants With Virologic Success Using the FDA-Defined Snapshot Analysis as Determined by the Achievement of HIV-1 RNA < 50 Copies/mL at Week 144
Time Frame: Week 144
Population: ITT Analysis Set
Measure: Number; unit: percentage of participants
Arm/Group | Stribild | ATV/r + FTC/TDF
Number analyzed (Participants) | 353 | 355
percentage of participants | 77.6 | 74.6

4. Secondary Outcome: The Percentage of Participants With Virologic Success Using the FDA-Defined Snapshot Analysis as Determined by the Achievement of HIV-1 RNA < 50 Copies/mL at Week 192
Time Frame: Week 192
Population: Week 192 modified intent-to-treat (MITT) Analysis Set: Participants in the ITT analysis set, excluding those who either 1) transferred to other Gilead-sponsored studies after completing their Week 144 Visit and before the lower limit of the Week 192 analysis window, or 2) prematurely discontinued study drug prior to the Week 144 Visit.
Measure: Number; unit: percentage of participants
Arm/Group | Stribild | ATV/r + FTC/TDF
Number analyzed (Participants) | 74 | 78
percentage of participants | 78.4 | 73.1

5. Secondary Outcome: The Percentage of Participants Achieving and Maintaining Confirmed HIV-1 RNA < 50 Copies/mL at Week 48 Using the FDA-defined Time to Loss of Virologic Response (TLOVR) Algorithm
Time Frame: Week 48
Population: ITT analysis set
Measure: Number; unit: percentage of participants
Arm/Group | Stribild | ATV/r + FTC/TDF
Number analyzed (Participants) | 353 | 355
percentage of participants | 86.1 | 84.8

6. Secondary Outcome: The Change From Baseline in Cluster Determinant 4 (CD4) Cell Count at Weeks 48, 96, 144, and 192
Description: Change = value of the relevant time point minus the baseline value
Time Frame: Baseline; Weeks 48, 96, 144, and 192
Population: ITT analysis set. The missing = excluded (M = E) method was used in which participants with missing data were excluded from analysis.
Measure: Mean (Standard Deviation); unit: cells/µL
Arm/Group | Stribild | ATV/r + FTC/TDF
Number analyzed (Participants) | 353 | 355
cells/µL
  Change at Wk 48 (Stribild, n=334; ATV/r, n=321) | 207 (164.2) | 211 (160.3)
  Change at Wk 96 (Stribild, n=317; ATV/r, n=315) | 256 (166.8) | 261 (188.0)
  Change at Wk 144 (Stribild, n=297; ATV/r, n=286) | 280 (159.8) | 293 (211.5)
  Change at Wk 192 (Stribild, n=69; ATV/r, n=72) | 338 (186.8) | 340 (224.2)

7. Secondary Outcome: The Percentage of Participants With HIV-1 RNA < 50 Copies/mL at Week 48
Time Frame: Week 48
Population: ITT analysis set. The missing = failure (M = F) method was used in which all missing data were considered as failure (HIV-1 RNA ≥ 50 copies/mL).
Measure: Number; unit: percentage of participants
Arm/Group | Stribild | ATV/r + FTC/TDF
Number analyzed (Participants) | 353 | 355
percentage of participants | 91.5 | 88.5

ADVERSE EVENTS:
Time Frame: Adverse events are reported for the double-blind treatment period of Stribild or ATV/r + Truvada up to 216 weeks plus 30 days.
Description: Safety Analysis Set: participants who were randomized into the study and received at least 1 dose of study drug
Arm/Group | Stribild | ATV/r + FTC/TDF
Serious Adverse Events (participants affected / at risk) | 58/353 | 62/355
Other Adverse Events (participants affected / at risk) | 326/353 | 326/355
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Stribild (N=353) | ATV/r + FTC/TDF (N=355)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1
Angina pectoris (Cardiac disorders) | 0 | 1
Myocardial infarction (Cardiac disorders) | 1 | 2
Congenital ureteric anomaly (Congenital, familial and genetic disorders) | 1 | 0
Iridocyclitis (Eye disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 4
Colitis (Gastrointestinal disorders) | 1 | 1
Constipation (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 0
Diverticulum (Gastrointestinal disorders) | 1 | 0
Erosive oesophagitis (Gastrointestinal disorders) | 1 | 0
Gastritis erosive (Gastrointestinal disorders) | 0 | 1
Haemorrhoids (Gastrointestinal disorders) | 1 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Large intestine perforation (Gastrointestinal disorders) | 0 | 1
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 1 | 0
Peptic ulcer haemorrhage (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1
Asthenia (General disorders) | 0 | 1
Chest pain (General disorders) | 1 | 1
Pyrexia (General disorders) | 1 | 0
Bile duct stone (Hepatobiliary disorders) | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 0 | 1
Drug hypersensitivity (Immune system disorders) | 1 | 0
Abscess limb (Infections and infestations) | 0 | 1
Abscess neck (Infections and infestations) | 0 | 1
Anal abscess (Infections and infestations) | 1 | 3
Appendicitis (Infections and infestations) | 3 | 1
Appendicitis perforated (Infections and infestations) | 1 | 0
Arthritis infective (Infections and infestations) | 1 | 0
Breast abscess (Infections and infestations) | 1 | 0
Bronchitis (Infections and infestations) | 1 | 0
Bronchopneumonia (Infections and infestations) | 0 | 1
Cellulitis (Infections and infestations) | 1 | 2
Device related infection (Infections and infestations) | 0 | 1
Ear infection (Infections and infestations) | 0 | 1
Epididymitis (Infections and infestations) | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 1
Gastroenteritis cryptosporidial (Infections and infestations) | 1 | 0
Gastrointestinal infection (Infections and infestations) | 0 | 1
Herpes zoster oticus (Infections and infestations) | 0 | 1
Impetigo (Infections and infestations) | 0 | 1
Incision site infection (Infections and infestations) | 0 | 1
Infectious colitis (Infections and infestations) | 1 | 0
Influenza (Infections and infestations) | 1 | 0
Lymphogranuloma venereum (Infections and infestations) | 1 | 0
Malaria (Infections and infestations) | 1 | 0
Malignant syphilis (Infections and infestations) | 1 | 0
Meningitis aseptic (Infections and infestations) | 0 | 1
Meningitis enteroviral (Infections and infestations) | 0 | 1
Meningitis viral (Infections and infestations) | 0 | 1
Orchitis (Infections and infestations) | 0 | 1
Osteomyelitis (Infections and infestations) | 1 | 1
Peritonitis (Infections and infestations) | 2 | 0
Pilonidal cyst (Infections and infestations) | 0 | 1
Pneumocystis jirovecii pneumonia (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 1 | 1
Pneumonia bacterial (Infections and infestations) | 1 | 0
Pneumonia streptococcal (Infections and infestations) | 1 | 0
Pyelonephritis acute (Infections and infestations) | 0 | 1
Respiratory syncytial virus infection (Infections and infestations) | 1 | 0
Salpingitis (Infections and infestations) | 1 | 0
Scrotal abscess (Infections and infestations) | 0 | 1
Secondary syphilis (Infections and infestations) | 1 | 0
Septic shock (Infections and infestations) | 0 | 2
Shigella infection (Infections and infestations) | 1 | 0
Staphylococcal infection (Infections and infestations) | 1 | 0
Tonsillitis (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 1 | 0
Viral infection (Infections and infestations) | 1 | 0
Alcohol poisoning (Injury, poisoning and procedural complications) | 1 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 1
Clavicle fracture (Injury, poisoning and procedural complications) | 1 | 0
Femur fracture (Injury, poisoning and procedural complications) | 1 | 0
Hand fracture (Injury, poisoning and procedural complications) | 0 | 1
Lower limb fracture (Injury, poisoning and procedural complications) | 0 | 1
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 | 0
Muscle rupture (Injury, poisoning and procedural complications) | 1 | 0
Muscle strain (Injury, poisoning and procedural complications) | 1 | 0
Overdose (Injury, poisoning and procedural complications) | 2 | 1
Post concussion syndrome (Injury, poisoning and procedural complications) | 1 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 1
Skull fractured base (Injury, poisoning and procedural complications) | 1 | 0
Toxicity to various agents (Injury, poisoning and procedural complications) | 1 | 2
Upper limb fracture (Injury, poisoning and procedural complications) | 1 | 1
Wrist fracture (Injury, poisoning and procedural complications) | 0 | 1
Blood creatine phosphokinase increased (Investigations) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Arthritis reactive (Musculoskeletal and connective tissue disorders) | 1 | 0
Foot deformity (Musculoskeletal and connective tissue disorders) | 0 | 1
Intervertebral disc displacement (Musculoskeletal and connective tissue disorders) | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 1
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 | 1
Anal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Anal squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Anogenital warts (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
B-cell lymphoma stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Burkitt's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Hodgkin's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Cervical radiculopathy (Nervous system disorders) | 1 | 0
Coma (Nervous system disorders) | 0 | 1
Convulsion (Nervous system disorders) | 2 | 0
Critical illness polyneuropathy (Nervous system disorders) | 0 | 1
Haemorrhage intracranial (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 0 | 1
Hypoaesthesia (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 1 | 1
Tension headache (Nervous system disorders) | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 1 | 0
VIIth nerve paralysis (Nervous system disorders) | 0 | 1
Alcohol withdrawal syndrome (Psychiatric disorders) | 1 | 1
Bipolar disorder (Psychiatric disorders) | 0 | 1
Depressed mood (Psychiatric disorders) | 0 | 1
Depression (Psychiatric disorders) | 3 | 1
Depressive symptom (Psychiatric disorders) | 0 | 1
Drug dependence (Psychiatric disorders) | 1 | 0
Major depression (Psychiatric disorders) | 1 | 0
Mania (Psychiatric disorders) | 0 | 1
Post-traumatic stress disorder (Psychiatric disorders) | 1 | 0
Schizophrenia (Psychiatric disorders) | 1 | 2
Substance abuse (Psychiatric disorders) | 0 | 1
Substance-induced psychotic disorder (Psychiatric disorders) | 1 | 0
Suicidal ideation (Psychiatric disorders) | 2 | 1
Suicide attempt (Psychiatric disorders) | 2 | 2
Hydronephrosis (Renal and urinary disorders) | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 1 | 0
Renal colic (Renal and urinary disorders) | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Respiratory depression (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Tonsillar hypertrophy (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Drug eruption (Skin and subcutaneous tissue disorders) | 0 | 1
Psoriasis (Skin and subcutaneous tissue disorders) | 0 | 1
Treatment noncompliance (Social circumstances) | 0 | 1
Orthostatic hypotension (Vascular disorders) | 0 | 1
Peripheral embolism (Vascular disorders) | 1 | 0
Thrombophlebitis (Vascular disorders) | 1 | 0
Venous thrombosis limb (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Stribild (N=353) | ATV/r + FTC/TDF (N=355)
Lymphadenopathy (Blood and lymphatic system disorders) | 23 | 16
Ocular icterus (Eye disorders) | 2 | 52
Abdominal pain (Gastrointestinal disorders) | 25 | 26
Constipation (Gastrointestinal disorders) | 20 | 14
Diarrhoea (Gastrointestinal disorders) | 99 | 121
Dyspepsia (Gastrointestinal disorders) | 13 | 19
Flatulence (Gastrointestinal disorders) | 16 | 32
Nausea (Gastrointestinal disorders) | 80 | 78
Vomiting (Gastrointestinal disorders) | 26 | 35
Fatigue (General disorders) | 60 | 60
Pyrexia (General disorders) | 23 | 22
Jaundice (Hepatobiliary disorders) | 0 | 34
Seasonal allergy (Immune system disorders) | 17 | 19
Bronchitis (Infections and infestations) | 47 | 42
Chlamydial infection (Infections and infestations) | 18 | 17
Folliculitis (Infections and infestations) | 19 | 22
Gastroenteritis (Infections and infestations) | 18 | 28
Herpes zoster (Infections and infestations) | 15 | 20
Influenza (Infections and infestations) | 31 | 24
Nasopharyngitis (Infections and infestations) | 53 | 57
Onychomycosis (Infections and infestations) | 21 | 13
Pharyngitis (Infections and infestations) | 23 | 18
Sinusitis (Infections and infestations) | 35 | 38
Syphilis (Infections and infestations) | 27 | 29
Upper respiratory tract infection (Infections and infestations) | 86 | 97
Urinary tract infection (Infections and infestations) | 18 | 20
Decreased appetite (Metabolism and nutrition disorders) | 14 | 19
Vitamin D deficiency (Metabolism and nutrition disorders) | 21 | 19
Arthralgia (Musculoskeletal and connective tissue disorders) | 35 | 32
Back pain (Musculoskeletal and connective tissue disorders) | 46 | 37
Pain in extremity (Musculoskeletal and connective tissue disorders) | 22 | 21
Anorectal human papilloma virus infection (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 21 | 12
Dizziness (Nervous system disorders) | 25 | 28
Headache (Nervous system disorders) | 67 | 55
Paraesthesia (Nervous system disorders) | 9 | 21
Anxiety (Psychiatric disorders) | 22 | 29
Depression (Psychiatric disorders) | 47 | 52
Insomnia (Psychiatric disorders) | 37 | 36
Cough (Respiratory, thoracic and mediastinal disorders) | 38 | 46
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 19 | 32
Night sweats (Skin and subcutaneous tissue disorders) | 10 | 18
Rash (Skin and subcutaneous tissue disorders) | 30 | 37
Hypertension (Vascular disorders) | 24 | 12

LIMITATIONS AND CAVEATS:
There were no limitations affecting the analysis or results.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years